CLINICAL TRIAL: NCT06080776
Title: A Phase III, Double-blind, Randomised Study of SH-1028 Tablets Versus Placebo as Adjuvant Therapy in Resected Stage II-IIIB Non-Small Cell Lung Cancer With Sensitizing EGFR Mutations
Brief Title: SH-1028 Tablets Versus Placebo as Adjuvant Therapy in Resected Stage II-IIIB NSCLC With Sensitizing EGFR Mutations
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHC013-III-02
Record Dates: First submitted 2023-08-08; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — SH-1028

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SH-1028 tablets (Experimental)
  Interventions: Drug: SH-1028 tablets
- Placebo SH-1028 tablets (Placebo Comparator)
  Interventions: Drug: Placebo SH-1028 tablets

INTERVENTIONS:
Drug: SH-1028 tablets — The initial dose of SH-1028 tablets is 200 mg once daily.
  Arms: SH-1028 tablets
Drug: Placebo SH-1028 tablets — Placebo SH-1028 tablets.
  Arms: Placebo SH-1028 tablets

SUMMARY:
To assess the efficacy and safety of SH-1028 tablets versus placebo in stage II-IIIB non-small cell lung cancer (NSCLC) patients with sensitizing epidermal growth factor receptor (EGFR) mutations, following complete tumor resection, with or without adjuvant chemotherapy.

DETAILED DESCRIPTION:
This is a Phase III, multi-center, double-blind, randomized study assessing the efficacy and safety of SH-1028 tablets (200 mg orally, once daily) versus placebo in stage II-IIIB NSCLC with sensitizing EGFR mutations, following complete tumor resection, with or without adjuvant chemotherapy (2~4 cycles of platinum-based doublet).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged at least 18 years, younger than 75 years.
* Histologically confirmed diagnosis of primary non-small lung cancer (NSCLC) on predominantly non-squamous histology.
* Before surgery or randomization, MRI or CT scan of the brain and bone scan must be done to exclude metastases.
* Complete resection (R0) and systematic lymphadenectomy are mandatory: all surgical margins must be negative for tumor, and there should be no extranodal invasion of the mediastinal lymph nodes or marginal lymph nodes.
* Patients with postoperative pathological confirmation of stage II, IIIA and IIIB (only T3N2M0) are eligible.
* Patients must harbor one of the two common sensitizing EGFR mutations (Ex19del, L858R), either alone or in combination with other EGFR mutations including T790M, the mutations should be confirmed by the central laboratory.
* Complete recovery from surgery and standard post-operative therapy (if applicable) at the time of randomization.
* A ECOG performance status equal to 0-1 with a minimum life expectancy of 12 weeks and no deterioration over the past 2 weeks.
* Adequate bone marrow reserve or organ function, as demonstrated by the following laboratory values (no corrective treatment allowed within one week before blood sampling):

  1. Absolute neutrophil count (ANC）≥1.5×10^9 /L
  2. Platelet count ≥100×10^9 /L
  3. Hemoglobin ≥90 g/L
  4. Alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or ≤ 5 × ULN in the presence of liver metastases
  5. Aspartate aminotransferase (AST) ≤ 2.5 × ULN if no demonstrable liver metastases or ≤ 5 × ULN in the presence of liver metastases
  6. Total bilirubin (TBL) ≤ 1.5 × ULN if no liver metastases or ≤ 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases
  7. Creatinine ≤ 1.5 × ULN concurrent with creatinine clearance ≥ 50 mL/min (measured or calculated by the Cockcroft-Gault equation); confirmation of creatinine clearance is only required when creatinine is ≤ 1.5×ULN
  8. Serum albumin (ALB) ≥28 g/L
  9. Coagulation function: International standardized ratio (INR) ≤1.5, activated partial thromboplastin time (APTT) ≤1.5×ULN
* Females of child-bearing potential should be using adequate contraceptive measures throughout the study, should not be breast feeding during the study and until 6 months after treatment, and must have a negative pregnancy test prior to start of dosing.
* Male patients should be willing to use barrier contraception during the study and until 6 months after treatment.
* Patients must sign and date written informed consent prior to admission to the study.

Exclusion Criteria:

* Patients with unresectable or metastatic lesions, residual lesions after surgery, or those who have had only segmentectomies or wedge resection.
* Giant mediastinal lymph node metastasis at a single station or mediastinal lymph node fusion into a cluster at multiple stations; lesions invade the heart, aorta, esophagus, or pulmonary veins; Carcinoma of superior lung sulci.
* Treatment with any of the following (except for standard platinum -based adjuvant chemotherapy), including any EGFR-TKI, systemic chemotherapy，immunotherapy, targeted therapy and anti-tumor traditional Chinese medicine therapy.
* Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug.
* The patient is currently using (or cannot discontinue at least 1 week before the first dose of study drug) a drug or herbal supplement known as a potent inhibitor or inducer of CYP3A4.
* Severe infections occurred within 4 weeks or active infections that received therapeutic intravenous or oral antibiotics within 2 weeks before the first dose.
* Any evidence of active infection (including hepatitis B, hepatitis C, and human immunodeficiency virus).
* Patients received continuous steroid therapy for more than 30 days within 30 days before the first dose; require long-term (≥30 days) steroid therapy; with acquired or congenital immunodeficiency diseases or have a history of organ transplantation.
* Severe or uncontrolled systemic diseases, including hypertension or diabetes.
* Any of the following cardiac criteria:

  1. Mean resting corrected QT interval (QTcF) > 470 msec obtained from 3 electrocardiograms (ECGs), using the Screening clinic's ECG machine and Fridericia's formula for QT interval correction.
  2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec).
  3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
  4. Left ventricular ejection fraction (LVEF) <50%.
* Receiving or requiring drugs known to prolong the QT interval or possibly cause tip torsion ventricular tachycardia during the study.
* History of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* History of any other malignant tumor within five years (except clinically cured cervical carcinoma in situ, basal cells or squamous epithelial skin cancer).
* Any seriously abnormal gastrointestinal function would affect uptake, transport and absorption of the drug, such as inability to swallow the study medication, refractory nausea and vomiting, previous significant bowel resection, Recurrent diarrhea, atrophic gastritis (age < 60 years), unhealed serious gastric diseases, Crohn's disease or ulcerative colitis.
* History of hypersensitivity to any active or inactive ingredient of SH-1028 or drug with a similar chemical structure or class to SH-1028.
* Any severe and uncontrolled ocular disease that may, in the Investigator's opinion, present a specific risk to the patient's safety.
* Participating in another clinical trial within 4 weeks before the first dose (excluding retrospective observational studies without intervention); within 5 half-lives of other study drugs.
* Hepatic encephalopathy, hepatorenal syndrome, or ≥Child-Pugh grade B cirrhosis.
* Lactating Women.
* Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival (DFS) assessed by Independent Review Committee (IRC) | From the time of randomization to the recurrence of tumor or death, through study completion, an average of 5 years
  Disease-free survival is defined as the time from randomization until the date of the recurrence of tumor or death. The primary endpoint of DFS was based on the assessment of IRC.

SECONDARY OUTCOMES:
Disease free survival (DFS) assessed by investigators | From the time of randomization to the recurrence of tumor or death, through study completion, an average of 5 years
  The secondary endpoint of DFS was based on the assessment of investigators.
DFS rate at 2, 3 and 5 years assessed by IRC | From the time of randomization to the recurrence of tumor or death, up to 5 years
  DFS rate at 2, 3 and 5 years is defined as the proportion of patients alive and disease free at 2, 3 and 5 years, respectively.
Overall survival (OS) | From the time of randomization to death, through study completion, an average of 5 years
  Overall survival is defined as the time from the date of randomization until death from any cause.
OS rate at 5 years | From the time of randomization to death, up to 5 years
  OS rate at 5 years is defined as the proportion of patients alive at 5 years.
Incidence rate of adverse events (AEs) | From the screening period to 28 days after treatment discontinuation
  AEs are assessed according to CTCAE v5.0.
Plasma concentrations of SH-1028 and its major metabolites | The specified time points of blood sampling, up to 36 weeks
  This is defined as the pharmacokinetics parameters derived from plasma concentrations of SH-1028 and its metabolites, Imp2 and Imp3.

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, Professor, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Daqiang Sun, Professor, Principal Investigator — Tianjin Chest Hospital, Tianjin, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China